CLINICAL TRIAL: NCT05166993
Title: Arterial Pressure Waveform Distortion: a New Dynamic Electronic Filter for Automatic Correction of Underdamping/Resonance Artifact. A Prospective Study
Brief Title: Dynamic Electronic Filter for Arterial Waveform Distortion
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Gianluca Villa, Professor, University of Florence
Other Study IDs: 10285
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Underdamping/Resonance Artifacts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: MostCareUp — Pressure transducers have been connected to the MostCareUp and the hemodynamic parameters compared as follows: no filter, electronic filter, no electronic filter plus Accudynamic (our reference system). Invasive pressure values have been then compared with the non-invasive ones.

SUMMARY:
Invasive blood pressure (IBP) is the gold standard for arterial pressure (AP) monitoring in critically ill patients. Nevertheless, IBP may be affected by underdamping/resonance artifacts, that eventually lead to AP overestimation. In these cases, when a pulse contour method is applied, wrong hemodynamic data are also delivered by the monitor. In order to overtake this issue, MostCareUp (a PCM powered by Pressure Recording Analytical Method, PRAM), has been implemented with a dynamic electronic filter (EFMC) that automatically corrects the resonant AP waveform.

In order to test the EFMC, the electronically corrected AP and the derived cardiac output were compared with respective raw data corrected with the Accudynamic, an adjustable damping device specifically manufactured for normalizing the pressure waveform (in our study: the reference method).

ELIGIBILITY:
Inclusion Criteria:

- ICU patients with invasive blood pressure (radial artery) affected by underdamping/resonance artifacts;

Exclusion Criteria:

- Arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to postoperative intensive care unit.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
The present study was aimed to test the MostCareUp electronic filter | 15 minutes
  To test the electronic filter comparing the electronically corrected arterial pressure and the derived cardiac output values with those corrected with the Accudynamic, a mechanical adjustable damping device commonly used in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Romagnoli, Prof, Study Director — University of Florence
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided